CLINICAL TRIAL: NCT00540293
Title: A Multicenter, Eight-Week Treatment, Single-Step Titration Open-Label Study Assessing The Percentage Of Korean Dyslipidemic Patients Achieving LDL Cholesterol Target With Atorvastatin Starting Doses Of 10 MG, 20 MG, And 40 MG.
Brief Title: Lipitor Korean Atorvastatin Goal Achievement Across Risk Levels Study
Acronym: AT GOAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2581157
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Results first posted 2009-06-26 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): this patient group consists of dyslipidemia patients with various CVD risk factors
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Prescription of 10/20/40mg dose atorvastatin based on the personal risk factor that is defined in the NCEP ATP III guideline in a single patient group

SUMMARY:
To evaluate the percentage of Korean dyslipidemic subjects in the total group and each cardiovascular risk group achieving LDL-C target as defined by NCEP ATP Ⅲ criteria at starting doses of 10mg, 20mg and 40mg of atorvastatin after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a Korean , dyslipidemic outpatient
2. Is eligible for LDL-lowering drug therapy at screening and baseline as determined by the following LDL-cholesterol (LDL-C) cut-off points defined by NCEP ATP Ⅲ: 2. 1 LDL-C ≥ 190 mg/dL for subjects with 0 or 1 CHD risk factor 2. 2 LDL-C ≥ 160 mg/dL for subjects with 2 or more CHD risk factors and 10 year risk < 10 % 2. 3 LDL-C ≥ 130 mg/dL for subjects with 2 or more CHD risk factors and 10 year risk 10-20 % 2. 4 LDL-C ≥ 100 mg/dL for subjects with documented CHD or CHD risk equivalents (10-year risk > 20 %)
3. Has LDL-C ≤ 220mg/dL at baseline 4. Has triglyceride level ≤ 600mg/dL at baseline

Exclusion Criteria:

1. Is pregnant or lactating
2. Has present myopathy or history of myopathy or has personal or familial history of hereditary muscular disorders or any history of rhabdomyolysis
3. Has history of intolerance or hypersensitivity to atorvastatin or other statins
4. Uncontrolled hypertension (i.e. moderate hypertension, sitting systolic BP ≥ 160mmHg and/or diastolic BP ≥ 100mmHg)
5. Has HbAlc > 10%
6. Has any severe disease of has had any major problem or surgical procedure within the 3 months prior to screening that is likely to jeopardize the planned termination of the study. (e.g., any carcinoma, coronary angioplasty, coronary artery bypass graft, cardiac infarct, severe or unstable angina pectoris)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- South Korea (10):
  - Pfizer Investigational Site, Daegu, Korea
  - Pfizer Investigational Site, Seoul, Korea
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Gyeonggi-do
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Kyunggi-do
  - Pfizer Investigational Site, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581157&StudyName=Lipitor%20Korean%20Atorvastatin%20Goal%20Achievement%20Across%20Risk%20Levels%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 20 centers in Korea
Pre-assignment Details: Participants who were on antilipidemic medications at the time of screening required a 6-week washout period prior to study treatment
Groups:
- Total Treatment Group (All Subjects Who Received Atorvastatin): this patient group consists of dyslipidemia patients with various cardiovascular diseases (CVD)risk factors
Period: Overall Study
Arm/Group | Total Treatment Group (All Subjects Who Received Atorvastatin)
Started | 425
Completed | 390
Not Completed | 35
Not completed — Adverse event related to study drug | 10
Not completed — Adverse event not related to study drug | 7
Not completed — Withdrawal by Subject | 6
Not completed — Protocol violation, & subject schedule | 12

BASELINE CHARACTERISTICS:
Arm/Group | Total Treatment Group (All Subjects Who Received Atorvastatin)
Number analyzed (Participants) | 425
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Females between 18 and 80 years | 62.9 (8.6)
  Males between 18 and 80 years | 58.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195
  Male | 230

OUTCOME MEASURES:

1. Secondary Outcome: Percent of Subjects in the Total Group and Each Cardiovascular Risk Group Achieving LDL-C Target After 4 Weeks of Treatment.
Description: LDL-C Responders by visit and by risk group - FAS
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: Percent subjects achieved LDL-C target
Groups:
- Total: N=425 (Total=sum of all risk groups)
- Low Risk: N=29 (Low Risk: Subjects with 0 or 1 CHD risk factor (who were assumed to have 10-year risk for CHD < 10%) or subjects with 2 or more CHD risk factors and 10-year risk for CHD < 10 %, e.g., subjects in Category 1 or 2.)
- Medium Risk: N=45 ( Medium Risk: Subjects with 2 or more CHD risk factors and 10-year risk for CHD 10-20 %, e.g., subjects in Category 3.)
- High Risk: N=351 (High Risk: Subjects with CHD, CHD risk equivalent or with 2 or more risk factors conferring a 10 year risk > 20 %, e.g., subjects in Category 4.)
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
Percent subjects achieved LDL-C target | 81.9 [77.9 to 85.5] | 85.7 [67.3 to 96.0] | 95.5 [84.5 to 99.4] | 79.9 [75.2 to 84.0]

2. Secondary Outcome: Changes in Lipid Parameters in Subjects in the Total Group and Each Cardiovascular Risk Group After 4 and 8 Weeks of Treatment
Description: Mean baseline, change and percent change from baseline in lipid parameters by risk group - FAS. HDL-C: high density lipoprotein-cholesterol; TC: total cholesterol; TG: triglyceride
Time Frame: Weeks 4 and 8
Measure: Mean (95% Confidence Interval); unit: mg/dL (ratio for Scalar)
Groups:
- Medium Risk: N=45 (Medium Risk: Subjects with 2 or more CHD risk factors and 10-year risk for CHD 10-20 %, e.g., subjects in Category 3.)
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
mg/dL (ratio for Scalar)
  LDL-C baseline | 151.7 [149.1 to 154.4] | 187.0 [179.8 to 194.1] | 160.6 [154.3 to 167.0] | 147.7 [144.9 to 150.5]
  LDL-C (week 4) | -63.5 [-66.2 to -60.8] | -73.8 [-82.7 to -64.8] | -65.1 [-73.5 to -56.7] | -62.4 [-65.4 to -59.4]
  LDL-C (week 8) | -65.3 [-68.0 to -62.5] | -77.6 [-88.3 to -66.9] | -64.2 [-72.4 to -56.0] | -64.4 [-67.4 to -61.4]
  HDL-C baseline | 48.3 [47.3 to 49.3] | 50.5 [47.4 to 53.7] | 48.0 [45.5 to 50.5] | 48.2 [47.0 to 49.3]
  HDL-C (week 4) | 0.1 [-0.7 to 0.9] | -0.8 [-3.6 to 2.0] | 3.3 [0.9 to 5.7] | -0.2 [-1.1 to 0.7]
  HDL-C (week 8) | 0.5 [-0.4 to 1.3] | 2.1 [-1.6 to 5.9] | 3.0 [0.9 to 5.1] | 0.0 [-1.0 to 1.0]
  Non-HDL-C baseline | 175.5 [172.5 to 178.5] | 209.9 [201.0 to 218.8] | 187.1 [179.9 to 194.4] | 171.1 [167.9 to 174.4]
  Non-HDL-C (week 4) | -69.4 [-72.3 to -66.5] | -75.4 [-87.8 to -63.1] | -71.3 [-80.2 to -62.5] | -68.6 [-71.8 to -65.4]
  Non-HDL-C (week 8) | -70.7 [-73.7 to -67.7] | -80.9 [-93.9 to -67.8] | -72.1 [-80.3 to -64.0] | -69.7 [-73.0 to -66.4]
  LDL-C/HDL-C ratio baseline | 3.2 [3.1 to 3.3] | 3.7 [3.4 to 4.0] | 3.4 [3.2 to 3.6] | 3.2 [3.1 to 3.3]
  LDL-C/HDL-C Ratio (Scalar) week 4 | -1.4 [-1.4 to -1.3] | -1.4 [-1.7 to -1.1] | -1.5 [-1.7 to -1.3] | -1.3 [-1.4 to -1.3]
  LDL-C/HDL-C Ratio (Scalar) week 8 | -1.4 [-1.5 to -1.3] | -1.6 [-1.9 to -1.2] | -1.5 [-1.7 to -1.3] | -1.4 [-1.5 to -1.3]
  TC baseline | 223.9 [220.8 to 227.0] | 262.3 [253.9 to 270.8] | 235.1 [228.0 to 242.3] | 219.3 [216.0 to 222.6]
  TC (week 4) | -69.4 [-72.4 to -66.4] | -78.2 [-89.3 to -67.1] | -68.0 [-77.2 to -58.8] | -68.8 [-72.2 to -65.5]
  TC (week 8) | -70.4 [-73.4 to -67.3] | -80.7 [-94.2 to -67.3] | -69.1 [-77.2 to -61.1] | -69.7 [-73.1 to -66.2]
  TG baseline | 154.1 [146.2 to 162.1] | 150.7 [128.6 to 172.8] | 152.3 [130.3 to 174.2] | 154.7 [145.6 to 163.7]
  TG (week 4) | -29.1 [-35.5 to -22.7] | -11.5 [-43.0 to 20.0] | -16.6 [-31.4 to -1.8] | -32.1 [-39.2 to -25.1]
  TG (week 8) | -29.3 [-37.9 to -20.7] | -20.9 [-51.3 to 9.5] | -18.5 [-36.3 to -0.7] | -31.4 [-41.3 to -21.5]

3. Secondary Outcome: Percent Changes From Baseline in Lipid Parameters in Subjects in the Total Group and Each Cardiovascular Risk Group After 4 and 8 Weeks of Treatment
Description: Mean percent changes from baseline in lipid parameters by risk group - FAS. HDL-C: high density lipoprotein-cholesterol; TC: total cholesterol; TG: triglyceride
Time Frame: weeks 4 and 8
Population: Laboratory Population: 10 subjects from FAS (n=425) were not included in Laboratory Population (n=415).
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
Percent
  LDL-C % change from baseline (week 4) | -40.9 [-42.3 to -39.5] | -39.5 [-44.1 to -35.0] | -39.6 [-43.8 to -35.5] | -41.2 [-42.8 to -39.6]
  LDL-C % change from baseline (week 8) | -42.0 [-43.4 to -40.7] | -41.2 [-46.6 to -35.8] | -39.3 [-43.5 to -35.1] | -42.5 [-44.0 to -41.0]
  HDL-C % change from baseline (week 4) | 1.7 [0.0 to 3.4] | -0.2 [-6.0 to 5.6] | 7.7 [2.3 to 13.1] | 1.1 [-0.8 to 2.9]
  HDL-C % change from baseline (week 8) | 2.6 [0.8 to 4.4] | 5.6 [-2.1 to 13.2] | 6.7 [2.3 to 11.1] | 1.8 [-0.2 to 3.9]
  Non-HDL-C % change from baseline (week 4) | -38.7 [-40.1 to -37.4] | -35.5 [-40.9 to -30.1] | -37.7 [-41.5 to -33.8] | -39.1 [-40.6 to -37.7]
  Non-HDL-C % change from baseline (week 8) | -39.4 [-40.7 to -38.1] | -38.2 [-44.1 to -32.2] | -38.3 [-42.1 to -34.5] | -39.7 [-41.1 to -38.2]
  LDL-C/HDL-C ratio % change from baseline (week 4) | -41.3 [-43.0 to -39.7] | -36.7 [-44.3 to -29.0] | -44.1 [-48.9 to -39.3] | -41.4 [-43.2 to -39.6]
  LDL-C/HDL-C ratio % change from baseline (week 8) | -42.6 [-44.3 to -40.9] | -41.6 [-49.5 to -33.7] | -42.9 [-48.0 to -37.7] | -42.6 [-44.5 to -40.8]
  TC % change from baseline (week 4) | -30.3 [-31.4 to -29.2] | -29.7 [-33.6 to -25.7] | -28.5 [-31.9 to -25.2] | -30.6 [-31.9 to -29.3]
  TC % change from baseline (week 8) | -30.7 [-31.9 to -29.6] | -30.4 [-35.2 to -25.5] | -29.2 [-32.3 to -26.2] | -31.0 [-32.2 to -29.7]
  TG % change from baseline (week 4) | -8.2 [-12.9 to -3.6] | 4.4 [-18.5 to 27.3] | -8.3 [-17.7 to 1.2] | -9.3 [-14.4 to -4.1]
  TG % change from baseline (week 8) | -9.8 [-14.9 to -4.8] | -6.3 [-27.0 to 14.5] | -7.0 [-20.4 to 6.4] | -10.5 [-16.2 to -4.8]

4. Secondary Outcome: Subjects Who Achieved LDL-C Target With no Titration of Atorvastatin and After One Step Titration of Atorvastatin.
Description: LDL-C responders at week 8 by titration status and risk groups - FAS, efficacy evaluation (EVAL), and FAS (no last observation carried forward, LOCF)
Time Frame: 8 weeks
Population: Laboratory Population: 10 subjects from FAS (n=425) were not included in Laboratory Population (n=415).
Measure: Number; unit: Participants
Groups:
- Low Risk: N=29(Low Risk: Subjects with 0 or 1 CHD risk factor (who were assumed to have 10-year risk for CHD < 10%) or subjects with 2 or more CHD risk factors and 10-year risk for CHD < 10 %, e.g., subjects in Category 1 or 2.)
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
Participants
  FAS population responders no titration | 339 | 24 | 41 | 274
  FAS population responders 1-step titration | 56 | 3 | 1 | 52
  EVAL population responders no titration | 305 | 22 | 39 | 244
  EVAL population responders 1-step titration | 53 | 3 | 1 | 49
  FAS population (no LOCF) no titration | 336 | 24 | 41 | 271
  FAS population (no LOCF) 1-step titration | 56 | 3 | 1 | 52

5. Secondary Outcome: Percent of Subjects Who Achieved LDL-C Target With no Titration of Atorvastatin and After One Step Titration of Atorvastatin.
Description: LDL-C responders at week 8 by titration status and risk groups - FAS, efficay evaluation (EVAL), and FAS (no last observation carried forward, LOCF)
Time Frame: 8 weeks
Population: Laboratory Population: 10 subjects from FAS (n=425) were not included in Laboratory Population (n=415).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
percentage of participants
  FAS population, no titration | 89.1 [85.3 to 92.2] | 95.8 [78.9 to 99.9] | 97.6 [87.1 to 99.9] | 87.2 [82.7 to 90.9]
  FAS population, 1-step titration | 82.1 [69.6 to 91.1] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0] | 80.8 [67.5 to 90.4]
  EVAL population, no titration | 91.1 [87.4 to 94.1] | 95.5 [77.2 to 99.9] | 97.4 [86.5 to 99.9] | 89.8 [85.2 to 93.3]
  EVAL population, 1-step titration | 83.0 [70.2 to 91.9] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0] | 81.6 [68.0 to 91.2]
  FAS population (no LOCF), no titration | 89.0 [85.1 to 92.1] | 95.8 [78.9 to 99.9] | 97.6 [87.1 to 99.9] | 87.1 [82.5 to 90.8]
  FAS population (no LOCF), 1-step titration | 82.1 [69.6 to 91.1] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0] | 80.8 [67.5 to 90.4]

6. Secondary Outcome: Change From Baseline in High Sensitive Circulating C-reactive Protein (Hs-CRP) After 4 and 8 Weeks of Treatment
Description: Median baseline, and change from baseline in hs-CRP by risk group - FAS
Time Frame: 4 and 8 weeks
Population: Laboratory Population: 10 subjects from FAS (n=425) were not included in Laboratory Population (n=415).
Measure: Median (95% Confidence Interval); unit: mg/dL
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
mg/dL
  Baseline | 0.108 [0.094 to 0.126] | 0.082 [0.060 to 0.112] | 0.075 [0.059 to 0.126] | 0.122 [0.102 to 0.137]
  Median change from baseline (week 4) | -0.008 [-0.014 to -0.005] | -0.008 [-0.028 to -0.001] | -0.002 [-0.014 to 0.023] | -0.010 [-0.018 to -0.005]
  Median change from baseline (week 8) | -0.015 [-0.021 to -0.009] | -0.011 [-0.034 to 0.018] | -0.001 [-0.021 to 0.010] | -0.018 [-0.027 to -0.010]

7. Primary Outcome: Percent of Subjects in the Total and Each Cardiovascular Risk Group Achieving Low Density Lipoprotein-cholesterol (LDL-C) Target After 8 Weeks of Treatment.
Description: LDL-C Responders by visit and by risk group - full analysis set (FAS)
Time Frame: Week 8
Population: N=number of subjects in the Full Analysis Set (FAS). Number of Participants Analyzed represents subjects with on-treatment lipid measures (missing values imputed by last observation carried forward)
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Groups:
- Total: N=425 (Total: sum of all risk groups)
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
Percentage of participants | 86.0 [82.3 to 89.2] | 92.9 [76.5 to 99.1] | 95.5 [84.5 to 99.4] | 84.3 [80.0 to 87.9]

8. Secondary Outcome: Percent Change From Baseline in High Sensitive Circulating C-reactive Protein (Hs-CRP) After 4 and 8 Weeks of Treatment
Description: Percent change from baseline in hs-CRP by risk group - FAS
Time Frame: 4 and 8 weeks
Population: Laboratory Population: 10 subjects from FAS (n=425) were not included in Laboratory Population (n=415).
Measure: Median (95% Confidence Interval); unit: percentage
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 415 | 28 | 44 | 343
percentage
  Median % change from baseline (week 4) | -12.346 [-21.429 to -4.651] | -13.941 [-35.055 to -1.923] | -2.553 [-22.951 to 25.926] | -16.197 [-24.182 to -4.523]
  Median % change from baseline (week 8) | -18.605 [-24.138 to -11.111] | -18.621 [-37.363 to 20.690] | -1.472 [-26.364 to 14.925] | -20.561 [-25.333 to -12.346]

9. Secondary Outcome: Changes From Baseline in Selected Inflammatory Markers After 8 Weeks of Treatment.
Description: Median baseline, and change from baseline in monocyte chemoattractant protein (MCP-1), interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha) by risk group - FAS
Time Frame: Baseline, and 8 weeks
Population: Laboratory Population: 17 subjects from FAS (n=425) were not included in Laboratory Population (n=408).
Measure: Median (95% Confidence Interval); unit: pg/dL
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 408 | 28 | 43 | 337
pg/dL
  MCP-1 baseline | 302.7 [295.0 to 311.7] | 305.2 [267.9 to 340.6] | 317.7 [294.2 to 386.4] | 301.6 [291.7 to 310.0]
  MCP-1 change from baseline (week 8) | 39.8 [21.3 to 66.7] | -15.0 [-61.4 to 45.9] | -22.4 [-102.9 to 42.6] | 59.4 [33.6 to 74.9]
  IL-6 baseline | 0.40 [0.40 to 0.50] | 0.30 [0.10 to 0.60] | 0.40 [0.30 to 0.80] | 0.50 [0.40 to 0.60]
  IL-6 change from baseline (week 8) | 0.00 [0.00 to 0.00] | 0.00 [-0.30 to 0.00] | -0.10 [-0.30 to 0.00] | 0.00 [0.00 to 0.00]
  TNF-alpha baseline | 0.10 [0.10 to 0.10] | 0.10 [0.10 to 0.30] | 0.20 [0.10 to 0.30] | 0.10 [0.10 to 0.10]
  TNF-alpha change from baseline (week 8) | 0.00 [0.00 to 0.00] | 0.00 [-0.10 to 0.00] | 0.00 [-0.10 to 0.00] | 0.00 [0.00 to 0.00]

10. Secondary Outcome: Percent Changes From Baseline in Selected Inflammatory Markers After 8 Weeks of Treatment.
Description: Percent changes from baseline in monocyte chemoattractant protein (MCP-1), interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha) by risk group - FAS
Time Frame: 8 weeks
Population: Laboratory Population: 17 subjects from FAS (n=425) were not included in Laboratory Population (n=408).
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Total | Low Risk | Medium Risk | High Risk
Number analyzed (Participants) | 408 | 28 | 43 | 337
percent
  MCP-1 % change (week 8) | 14.0 [7.8 to 22.3] | -5.6 [-18.6 to 18.7] | -8.0 [-34.2 to 21.4] | 18.2 [11.1 to 24.7]
  IL-6 % change (week 8) | 0.00 [0.00 to 0.00] | 0.00 [-50.00 to 0.00] | -12.50 [-45.45 to 25.00] | 0.00 [0.00 to 0.00]
  TNF-alpha % change (week 8) | 0.00 [0.00 to 0.00] | 0.00 [-50.00 to 0.00] | 0.00 [-42.86 to 0.00] | 0.00 [0.00 to 0.00]

ADVERSE EVENTS:
Arm/Group | Total Treatment Group (All Subjects Who Received Atorvastatin)
Serious Adverse Events (participants affected / at risk) | 3
Other Adverse Events (participants affected / at risk) | 14
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Total Treatment Group (All Subjects Who Received Atorvastatin)
Wrist fracture (Injury, poisoning and procedural complications) | 1/425
Cerabral infarction (Nervous system disorders) | 2/425
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Total Treatment Group (All Subjects Who Received Atorvastatin)
Nasopharyngitis (Infections and infestations) | 8/425
Headache (Nervous system disorders) | 6/425

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.